CLINICAL TRIAL: NCT04026321
Title: A Double-blind, Single-dose Escalation Study of SQ-001 Infusion at a Single Center to Characterize the PK Profiles of Major Sentinel Compounds, Astragaloside IV, Calycosin 7-O-beta-glucopyranoside, and Lobetyolin in the Plasma of Healthy Adult Volunteers in the United States
Brief Title: Single-dose Escalation Study of SQ-001 Infusion to Characterize the PK Profiles of Major Sentinel Compounds in Healthy Adult Volunteers in US
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Collaborators: Palm Beach CRO (Unknown); Keystone Bioanalytical, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LV-SQ001-01
Record Dates: First submitted 2019-07-14; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Solid Tumor Refractory to Standard Therapy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SQ-001 125mL/day (Experimental)
  Interventions: Drug: SQ001 125mL/day
- SQ-001 250mL/day (Experimental)
  Interventions: Drug: SQ001 250mL/day
- SQ-001 500mL/day (Experimental)
  Interventions: Drug: SQ001 500mL/day
- SQ-001 625mL/day (Experimental)
  Interventions: Drug: SQ001 625mL/day
- saline(0.9% NaCl injection) (Placebo Comparator)
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: SQ001 125mL/day — SQ001 125mL/day will be administered by intravenous route at a rate of 3 mL/minute
  Arms: SQ-001 125mL/day
Drug: SQ001 250mL/day — SQ001 250mL/day will be administered by intravenous route at a rate of 3 mL/minute
  Arms: SQ-001 250mL/day
Drug: SQ001 500mL/day — SQ001 500mL/day will be administered by intravenous route at a rate of 3 mL/minute
  Arms: SQ-001 500mL/day
Drug: SQ001 625mL/day — SQ001 625mL/day will be administered by intravenous route at a rate of 3 mL/minute
  Arms: SQ-001 625mL/day
Drug: Saline 0.9% — Saline 0.9% will be administered by intravenous route at a rate of 3 mL/minute
  Arms: saline(0.9% NaCl injection)

SUMMARY:
This is a single-center, double-blind, single-dose escalation study in healthy volunteers.

DETAILED DESCRIPTION:
This is a single-center, double-blind, single-dose escalation study in healthy volunteers consisting of a 14-day Screening Period, 1-day Predose period, a 2-day Dosing and Evaluation Period, and a 5-day Follow-up Period, with a single Follow-up call scheduled on Day 7 ± 1. Subjects will be confined to the study site for up to 3 days (admitted on Day -1 and discharged on Day 2 or 3, depending on cohort) and will be monitored for adverse events (AEs) and dose limiting toxicities (DLT) during the Dosing, Evaluation and Follow-up Periods. Subjects will also be monitored for concomitant medications and use of rescue medications throughout the study.

Subjects will be allocated 1:4 to receive an infusion of saline control (0.9% saline for injection) or Shenqi Fuzheng Injection(SQ-001) continuously for about 1-4 hours. SQ 001 will be administered by intravenous route at a rate of 3 mL/min to one of four final dosages: Cohort 1 (125 mL/day/person), Cohort 2 (250 mL/day/person), Cohort 3 (500 mL/day/person), and Cohort 4 (625 mL/day/person). Each cohort will be enrolled sequentially. Per cohort, three subjects will be dosed initially on Day 1 and observed for 24 hours. If there are no observed AEs that meet the criteria under Stopping Rules, the remaining 7 subjects/cohort will be dosed. Dose escalation to the next higher dose will be based on the observation of results in safety and degree of AEs from the previous cohort and discussion between the Investigator and Sponsor.

A maximum 17 PK samples will be collected over the course of the study in each cohort. The PK sampling time points will be grouped as (a) pre-infusion; (b) intra-infusion; (c) completion of infusion; and (d) post-infusion. See Table 10 for plasma PK sampling times. The last PK sample will be collected 24 hours after the end of infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be medically documented as healthy at the time of screening as determined by their medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory tests, unless the Investigator considers an abnormality to be clinically irrelevant.
2. Subjects must be within 18 to 65 years old and not currently using tobacco products.
3. Subjects must have a BMI within 18 to 32 kg/m2.
4. Females

   1. Surgically sterilized (e.g., hysterectomy or bilateral oophorectomy) for at least 6 months prior to screening or postmenopausal (postmenopausal women must have no menstrual bleeding for at least 1 year prior to screening and menopause will be confirmed by a plasma FSH level of >30 IU/L) or
   2. Women of child-bearing potential must be non-lactating and agree to use a highly effective acceptable form of birth control such as surgical sterilization (e.g., tubal ligation), or total abstinence from sexual intercourse with the opposite sex, or established hormonal birth control (e.g. oral, implant or injection) plus a barrier method, or a double barrier method (e.g. intrauterine device plus condom or spermicidal gel plus condom or diaphragm plus condom) from 14 days prior to dosing until 30 days after dosing.
   3. Women with a negative serum pregnancy test (βhCG assay) at screening and at Day -1 (urine)
   4. For non-sexually active females, abstinence may be regarded as an adequate method of birth control, but if the subject becomes sexually active during the study, she must use adequate birth control as defined above for the remainder of the study.
5. Males Must be willing to use highly effective forms of acceptable birth control (e.g., vasectomy, total abstinence from sexual intercourse with the opposite sex, sexual intercourse with a woman who is not of childbearing potential) from Day 1 dosing to Day 90 after dose.
6. Subjects must be able to comply with the study and follow-up procedures.
7. Subjects must provide a signed informed consent to participate in the study.
8. Subjects must not have participated in any clinical trial within 30 days.

Exclusion Criteria:

1. Any condition preventing reliable phlebotomy or infusion from the cubital fossa.
2. Documented history of clinically significant unstable medical illness.
3. History of clinically significant drug, food, or environmental allergy.
4. Subjects with any uncontrolled medical condition deemed clinically significant by an Investigator.
5. Clinically significant safety laboratory, 12-lead ECG, or vital sign abnormalities during screening or Day -1 that would place the subject at undue risk based on the Investigator's opinion, including but not limited to:

   1. History of cardiac conditions that might give a higher risk of an increase in heart rate
   2. Fridericia's corrected QT interval (QTcF) interval of >450 msec on 12-lead ECG
   3. Alanine aminotransferase (ALT) >1.2 × upper limit of normal (ULN), aspartate aminotransferase (AST) >1.2 × ULN
   4. Blood urea nitrogen (BUN) or serum creatinine >1.2 × ULN
6. Subjects who are positive for HIV, HBV, and/or HCV.
7. Subjects who have used prescription drugs, over-the-counter drugs, or herbal remedies within 14 days before Day 1 of study medication dosing.
8. Women who are pregnant or breast feeding.
9. Subjects who participated in a clinical trial within 30 days prior to Day 1 study medication dosing.
10. Subjects with any condition that, in the judgment of the Principal Investigator, would place a subject at undue risk, or potentially compromise the results or interpretation of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
The maximum observed concentrations (Cmax)(ng/mL) | On 1 and 2 days (dosing day and the following evaluation day)
  To compare the Cmax of 3 major representative (sentinel) compounds astragaloside IV, calycosin 7-O-β-glucopyranoside, and lobetyolin in different experimental arms
Time to reach Cmax (Tmax)(h) | On 1 and 2 days (dosing day and the following evaluation day)
  To compare the Tmax of 3 major representative (sentinel) compounds astragaloside IV, calycosin 7-O-β-glucopyranoside, and lobetyolin in different experimental arms
Area under the concentration-time curve (AUC)(ng·h/mL) | On 1 and 2 days (dosing day and the following evaluation day)
  To compare the AUC of 3 major representative (sentinel) compounds astragaloside IV, calycosin 7-O-β-glucopyranoside, and lobetyolin in different experimental arms
Elimination half-life (T1/2)(h) | On 1 and 2 days (dosing day and the following evaluation day)
  To compare the Cmax of 3 major representative (sentinel) compounds astragaloside IV, calycosin 7-O-β-glucopyranoside, and lobetyolin in different experimental arms
Apparent clearance (CL)(mL/min/kg) | On 1 and 2 days (dosing day and the following evaluation day)
  To compare the CL of 3 major representative (sentinel) compounds astragaloside IV, calycosin 7-O-β-glucopyranoside, and lobetyolinin different experimental arms
Volume of distribution at steady state (Vdss)(L/kg) | On 1 and 2 days (dosing day and the following evaluation day)
  To compare the Vdss of 3 major representative (sentinel) compounds astragaloside IV, calycosin 7-O-β-glucopyranoside, and lobetyolinin different experimental arms

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events | From predose to up 5 days following the dosing and evaluation period
  Incidence of treatment-related adverse events as assessed by CTCAE v4.03
Frequency of treatment-related adverse events | From predose to up to 5 days following the dosing and evaluation period
  Frequency of treatment-related adverse events as assessed by CTCAE v4.03
Grade of treatment-related adverse events | From predose to up to 5 days following the dosing and evaluation period
  Grade of treatment-related adverse events as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Maria I. Bermudez, MD.CPI, Principal Investigator — Clinical Pharmacology of Miami, Inc.
Locations (1):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No